CLINICAL TRIAL: NCT00418873
Title: A Multi-centre Comparative Study to Evaluate the Anti-aggression Effect and Safety of Zotepine Versus Risperidone in Aggressive Schizophrenic Patients of Acute Ward
Brief Title: Zotepine Versus Risperidone in Aggressive Schizophrenic Patients of Acute Ward
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped due to difficulty in patient enrollment
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Director, Astellas Pharma Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPRIS-0601-TW
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; zotepine; risperidone; second generation antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — zotepine; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Zotepine (Experimental)
  Interventions: Drug: Zotepine
- 2. Risperidone (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Zotepine — Oral
  Other Names: Lodopin®; Zoleptil®; Nipolept®
  Arms: 1. Zotepine
Drug: Risperidone — Oral
  Other Names: Risperdal®
  Arms: 2. Risperidone

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability of zotepine versus Risperidone in aggressive schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years, male or female
* In-patients suffering from schizophrenia according to DSM-IV diagnostic criteria with PANSS total score of greater than or equal to 60.
* Patients with PANSS-EC total score of greater than or equal to 14 and with at least one PANSS-EC symptom score greater than or equal to 4

Exclusion Criteria:

* Patients with history of seizure or with alcohol or substance abuse in the last 6 months
* Diabetes, Parkinson's disease or phaeochromocytoma
* Patients with hypertension and current use of antihypertensive agents
* Women who are pregnant, lactating or intend to become pregnant during the study period
* Poor response to two different antipsychotics in full dose and full course or use of clozapine previously
* Renal, hepatic, haematologic disease or other conditions may not suitable for the study based on investigator's evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in aggression behavior assessed using the Positive and Negative Syndrome Scale Excited Component (PANSS-EC) score. | 6 Weeks

SECONDARY OUTCOMES:
Change from baseline on the total score of Positive and Negative Syndrome Scale | 6 Weeks
Change from baseline on Clinical Global Impression (CGI) | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Jer Tsai, Principal Investigator — Taipei City Hospital
Locations (3):
- Taiwan (3):
  - Bali, Taipei
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Chan HY, Lin AS, Chen KP, Cheng JS, Chen YY, Tsai CJ. An open-label, randomized, controlled trial of zotepine and risperidone for acutely ill, hospitalized, schizophrenic patients with symptoms of agitation. J Clin Psychopharmacol. 2013 Dec;33(6):747-52. doi: 10.1097/JCP.0b013e31829e8168. PMID 24100785